CLINICAL TRIAL: NCT02658305
Title: Transoral Versus Transbuccal Placement of Bicortical Screws During Orthognathic Surgery
Status: Completed | Type: Observational
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Johan Abeloos, Maxillofacial surgeon, Head of Department, AZ Sint-Jan AV
Other Study IDs: B049201525558
Record Dates: First submitted 2016-01-11; First posted 2016-01-18 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Prognathism; Retrognathia; Jaw Abnormalities
Keywords: transoral approach; transbuccal approach; postoperative complications
MeSH Terms: conditions — Prognathism; Retrognathia; Jaw Abnormalities; Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- transoral group: orthognathic patients that were treated with a transoral surgical approach
- transbuccal group: orthognathic patients that were treated with a transbuccal surgical approach

SUMMARY:
Bicortical screws have been widely used for mandibular osteosynthesis during orthognathic surgery.Transoral placement of bicortical screws is a rigid fixation method in orthognathic surgery, which is less often used.

The aim of this study was to compare postoperative outcome of transoral versus transbuccal bicortical screw placement during orthognathic surgery.

This study comprises an academic, retrospective, monocentric study in which the charts of orthognathic patients operated between January 2010 and December 2012 were retrospectively reviewed. Postoperative complications were registered. Demographic, dental and surgical parameters are examined as potential risk factors for the occurence of postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* patients of all ages
* patients of all genders
* patients who had undergone a bimaxillary osteotomy, a bilateral sagittal split ramus osteotomy (BSSO), a BSSO with a chin osteotomy or a trimaxillary osteotomy

Exclusion Criteria:

* patients where cement had been used at the osteotomy sites
* patients who had undergone a multisegmented mandibular osteotomy
* patients who had undergone an osteosynthesis with plates
* patients where the postoperative orthopantomogram was unavailable
* patients where data regarding the type of screw placement was unavailable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All orthognathic patients operated in the lower jaw between January 2010 and December 2012 at the Department of Oral and Maxillofacial Surgery, General Hospital Saint-John Bruges, Belgium
Sampling Method: Non-Probability Sample
Enrollment: 509 (Actual)
Dates: Start 2014-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Postoperative complications (rate of screw removal and/or infection) | within 4 weeks postoperative

SECONDARY OUTCOMES:
The value of demographic, dental and surgical parameters as potential risk factors for the occurence of postoperative complications | within 4 weeks postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Johan Abeloos, MD, Principal Investigator — Department of Oral and Maxillofacial Surgery, General Hospital Saint-John Bruges, Bruges, Belgium
Locations (1):
- General Hospital Saint-John Bruges, Bruges, Belgium

IPD SHARING:
Plan to Share IPD: No